CLINICAL TRIAL: NCT07032727
Title: Olutasidenib Combined With Co-targeted Therapy in Relapsed or Refractory IDH1-mutated Myeloid Malignancies Harboring Activated Signaling Pathway Mutations
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0520; NCI-2025-04331 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-06-16; First posted 2025-06-24 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-10

CONDITIONS: Targeted Therapy; IDH1-Mutated Malignancies; Mutations
MeSH Terms: interventions — olutasidenib; Cladribine; venetoclax; gilteritinib; ruxolitinib; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Arm 1A Safety Lead-In/Expansion: (Experimental): Treatment with Olutasidenib + Cladribine + Cytarabine
  Interventions: Drug: Olutasidenib; Drug: Cladribine (CLAD); Drug: Cytarabine
- Arm 1B Expansion (Experimental): Treatment with Olutasidenib + Cladribine + Cytarabine + Venetoclax
  Interventions: Drug: Olutasidenib; Drug: Cladribine (CLAD); Drug: Venetoclax; Drug: Cytarabine
- Arm 2A Safety Lead-In/Expansion (Experimental): Treatment with Olutasidenib + Gilteritnib
  Interventions: Drug: Olutasidenib; Drug: Gilteritinib
- Arm 2B Expansion (Experimental): Treatment with Olutasidenib + Gilteritnib + Venetoclax
  Interventions: Drug: Olutasidenib; Drug: Venetoclax; Drug: Gilteritinib
- Arm 3A Safety Lead-In/Expansion: (Experimental): Treatment with Olutasidenib + Ruxolitinib
  Interventions: Drug: Olutasidenib; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Olutasidenib — Given by po
Drug: Cladribine (CLAD) — Given by IV
  Arms: Arm 1A Safety Lead-In/Expansion:; Arm 1B Expansion
Drug: Venetoclax — Given by po
  Arms: Arm 1B Expansion; Arm 2B Expansion
Drug: Gilteritinib — Given by po
  Arms: Arm 2A Safety Lead-In/Expansion; Arm 2B Expansion
Drug: Ruxolitinib — Given by po
  Arms: Arm 3A Safety Lead-In/Expansion:
Drug: Cytarabine — Given SQ
  Arms: Arm 1A Safety Lead-In/Expansion:; Arm 1B Expansion

SUMMARY:
To learn about the safety and tolerability of study drug combinations in patients with relapsed/refractory, IDH1-mutated myeloid malignancies with a co-signaling mutation.

DETAILED DESCRIPTION:
Primary Objectives

1. To determine the safety and tolerability of olutasidenib in combination with cladribine + LDAC ± venetoclax (Arm 1), gilteritinib ± venetoclax (Arm 2), and ruxolitinib (Arm 3) for patients with relapsed/refractory IDH1-mutated myeloid malignancies with a co-signaling mutation.
2. To quantify the composite complete remission rate (CRc; CR + CRh + CRi) in patients with relapsed/refractory IDH1-mutated myeloid malignancies with a co-signaling mutation treated with olutasidenib in combination with cladribine + LDAC ± venetoclax (Arm 1), gilteritinib ± venetoclax (Arm 2), and ruxolitinib (Arm3).

Secondary Objectives

1. To determine overall survival (OS), event free survival (EFS), and duration of response (DOR) with olutasidenib in combination with a co-targeting chemotherapeutic agent.
2. To determine the overall response rate (ORR; CR + CRh + CRi + MLFS + PR) of olutasidenib in combination with a co-targeting chemotherapeutic agent.
3. To evaluate occurrence of measurable residual disease (MRD) negative status by multiparameter flow cytometry and molecular evaluation by polymerase chain reaction (PCR) and next generation sequencing (NGS)-based assays (e.g. IDH1 and FLT3 if applicable).
4. To characterize the pharmacokinetic (PK) profiles of olutasidenib and venetoclax in plasma samples.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years.
2. Participants with a diagnosis of relapsed and/or refractory AML (including biphenotypic or bilineage leukemia including a myeloid component) OR high-risk MDS, MPN, or MDS/MPN (defined as ≥10% blasts on peripheral flow cytometry or bone marrow biopsy).
3. Participants must have a documented IDH1 mutation.
4. Participants must also have a documented co-signaling mutation in one or more of the following: KRAS, NRAS, PTPN11, CBL, NF1, FLT3-ITD, FLT3-TKD, KIT, JAK2, MPL, CALR, CSF3R.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2.
6. Adequate renal function with estimated GFR ≥ 30 by the 2021 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI).
7. Adequate hepatic function, defined as direct bilirubin ≤ 2x upper limit of normal (ULN) and AST and ALT ≤ 3x ULN unless the increase is due to Gilbert's disease or leukemic involvement, in which case direct bilirubin, AST, and ALT ≤ 5x ULN will be considered eligible.
8. The interval from prior treatment to time of initiation will be at least 14 days OR five half-lives for both cytotoxic and non-cytotoxic (e.g. immunotherapy agent(s)). Oral hydroxyurea and/or cytarabine (up to 2g/m2) is allowed for participants with rapidly proliferative disease prior tothe start and during the first two cycles of therapy, for clinical benefit and after discussion with the PI. Continuation of concurrent intrathecal therapy for controlled CNS disease is permitted.
9. Ability to understand and the willingness to sign an informed consent document.

Exclusion Criteria

1. Participants who have received prior olutasidenib (Rezlidhiai, previously FT-2102).
2. Participants with translocation t(15;17) or acute promyelocytic leukemia (French-American British (FAB) class M3-AML).
3. Participants with any concurrent uncontrolled clinically significant medical condition, including life threatening infection, which could place the patient at unacceptable risk of study treatment.
4. Participants with any uncontrolled psychiatric illness that would limit compliance with study requirements.
5. Participants with a New York Heart Association (NYHA) Functional Classification of III or IV.

   • Participants with active graft-versus-host-disease (GVHD) status post stem cell transplant (Participants without active GVHD on phototherapy for chronic skin GVHD are permitted after discussion with the PI). Participants must have discontinued calcineurin inhibitors at least 4 weeks prior to the start of study treatment.
6. Participants with active, uncontrolled CNS leukemia.
7. Participants with any severe gastrointestinal or metabolic condition which could interfere with the absorption of oral study medications.
8. Known active hepatitis B (HBV), hepatitis C (HCV), or human immunodeficiency virus (HIV) infection. For participants with evidence of chronic HBV or HIV infection, the HBV or HIV viral load must be undetectable, respectively. For participants with a history of HCV, it must be treated and cured with an undetectable HCV viral load.
9. Participant has white blood cell count >25 x 109/L (Note: Hydroxyurea and cytarabine are permitted to mean this criterion).
10. The effects of the study drug on the developing human fetus or transmission through breast feeding are unknown. Therefore, nursing women and women with a positive urine pregnancy test and excluded. Additionally, women of child-bearing potential (WOCBP) and men who are sexually active with WOCBP who are not willing to maintain adequate contraception are excluded.

    a. WOCBP includes all female participants between the onset of menses (as early as 8 years of age) to 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following: i. Postmenopausal (no menses in greater than or equal to 12 consecutive months).

    ii. History of hysterectomy or bilateral salpingo-oophorectomy. iii. Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).

    iv. History of bilateral tubal ligation or another surgical sterilization procedure.

    b. Approved methods of birth control are as follows: hormonal contraception (i.e. birth control pills, injection, transdermal patch, vaginal ring, hormonal implant), intrauterine device (IUD), tubal ligation or hysterectomy, subject/partner post-vasectomy, double barrier methods (e.g. condom in combination with spermicide). Abstinence for the duration of the trial and drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform the treating physician immediately.

    c. Adequate contraception must be maintained from initiation of the study drug until 90 days after the last dose of the study drug.
11. History of an allergic reaction to venetoclax, gilteritinib, ruxolitinib, cladribine, or cytarabine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org